CLINICAL TRIAL: NCT03474705
Title: Clinical Outcomes, Muscle Stiffness and Creep, and Central Pain Mechanisms Are Improved After Eccentric Training in Female Computer Users With Chronic Neck/Shoulder Pain
Brief Title: Clinical Outcomes, Viscoelastic Properties and Central Pain Mechanisms After Eccentric Training in Neck/Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Alberto Marcos Heredia-Rizo, Assistant Professor, University of Seville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMHRizo
Record Dates: First submitted 2018-03-05; First posted 2018-03-22 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Neck Pain; Work-related Injury; Shoulder Pain
Keywords: Clinical Pain; Hyperalgesia; Intervention; Musculoskeletal disorders; Computer Work; Strength Training
MeSH Terms: conditions — Neck Pain; Shoulder Pain; Hyperalgesia; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eccentric Training Group (Experimental): Eccentric training of the upper trapezius muscles. The intervention will consist of ten sessions of 25-30 minutes (twice a week over 5 consecutive weeks) of eccentric exercises of the shoulder muscles, as neural activation increases after 4 weeks of eccentric training. The total duration of the intervention will be 2 hours and a half.
  Interventions: Device: Eccentric Training Protocol

INTERVENTIONS:
Device: Eccentric Training Protocol — A custom-built dynamic shoulder dynamometer (Aalborg University, Aalborg, Denmark) will be used. Participants will be seated with back support and no feet support. The maximal voluntary contraction (MVC) of the painful side will be assessed. Sessions will start with a 5-min warm-up. After that, participants will sit in the dynamometer, and the range of shoulder elevation (highest and lowest vertical position) will be measured for the affected side. During training, subjects will have to counteract a dynamometer vertical force from the highest to the lowest shoulder position at a force equal to 60% (training sessions 1-3), 70% (training sessions 4-6), and 80% (training sessions 7-10) of the MVC recorded during baseline. Three bouts of 10 repetitions (sessions 1-3), 8 repetitions (sessions 4-6) and 6 repetitions (sessions 7-10) will be performed, with a 3-second rest between contractions and a 2-minute break between bouts.

SUMMARY:
Objectives: The aims are to 1) evaluate the clinical impact of eccentric training in female computer users with chronic NSP, 2) compare pressure hyperalgesia, temporal summation of pain (TSP), and conditioned pain modulation (CPM) in female office workers with and without NSP, and 3) assess changes in central pain responses after training.

Methods: In part A, twenty office workers with NSP will be compared with 20 healthy controls. In part B, the NSP group will undergo a 5-week eccentric training program. Participants will report their pain intensity, and complete the Neck Disability Index, and the Disabilities of the Arm, Shoulder and Hand questionnaire. Pressure pain thresholds (PPTs) will be assessed over the neck and forearm. Cuff algometry will identify pain detection (PDT) and tolerance thresholds (PTT). TSP will be evaluated by visual analogue scale pain scores during 10 repetitive cuff stimulations. CPM will be calculated as the difference in PDT with and without a conditioning painful stimulus. Outcomes will be measured at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Neck / shoulder pain has to last more than 12 weeks', with an average score higher than 2 on a 11-point Numeric Pain Rating Scale within the last 24 hours and during the week before data collection.
* All subjects will have to work for a minimum of four hours per day using a computer, should speak and understand English, and could not be involved in regular strength training of the neck/upper extremities

Exclusion Criteria:

* previous whiplash; a history of neurological or mental illnesses; consumption of pain killers within the last 24 hours; drug addiction, defined as the use of cannabis, opioids or other drugs; fibromyalgia; previous cervical spine or upper limb surgery; carpal tunnel syndrome; concomitant injury or pain from the lumbar spine; and heart diseases or hypertension.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity, assessed by a 11-point Numeric Pain Rating Scale (NPRS) | Change from Baseline to Pain Level after a two-week intervention protocol
  It will be measured the worst pain within the last 24 hours and the average pain intensity during the previous week
Upper limb function, assessed by the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Change from Baseline to Upper extremity Disability Level after a two-week intervention protocol
  The DASH questionnaire is the most recommended scale to assess individuals with shoulder disorders
Neck disability, assessed by the Neck Disability Index (NDI) | Change from Baseline to Neck Disability Level after a two-week intervention protocol
  The NDI is a valid and reliable tool, frequently used to assess functionality in workplace interventions

SECONDARY OUTCOMES:
Pressure Pain Threshold, assessed by Manual Pressure Algometry | Change from Baseline to after a two-week intervention protocol
  A handheld electronic pressure algometer with a 1-cm2 contact probe will be used. Pressure pain thresholds (PPTs), as the minimum necessary pressure force to evoke pain, will be assessed bilaterally over the middle point of the upper trapezius muscle belly, and the muscle bellies of the extensor carpi radialis brevis and the extensor carpi ulnaris. A 30-second break will be used between assessments to prevent bruising, and an average of the two measures over each site will be calculated for the statistical analysis. Pressure algometry is reliable in healthy individuals, and in neck pain.
Cuff Algometry | Change from Baseline to after a two-week intervention protocol
  A computer-controlled cuff-algometer (Aalborg University, Aalborg, Denmark) will be used to evaluate distal hyperalgesia at the lower legs by means of pain detection (PDT) and tolerance threshold (PTT). A single 13-cm-wide cuff (VBM, Sulz am Neckar, Germany) will be wrapped around the gastrocnemius muscles, at the level with the maximum circumference, on both sides. The cuff pressure will be increased by 1 kPa/s, with the maximal pressure set up at 100 kPa. Participants will be told to rate their pain intensity on a 10-cm electronic Visual Analogue Scale (VAS), and to press a button to release the cuff inflation when the pain was unbearable (PTT). PDT will be considered as the pressure corresponding to the first VAS rating more than 1 cm. This protocol is highly reliable and an examiner-independent procedure.
Temporal Summation of Pain (TPS) | Change from Baseline to after a two-week intervention protocol
  TSP will be collected from the painful/most painful side, and the same side matched on dominance for controls. Ten consecutive cuff pressure stimuli (1-second duration, 1-second break interval) will be delivered by inflating the cuff chamber at the same intensity than the PTT . During intervals, a non-painful pressure of 1 kPa will be applied. Participants will have to continuously rate their pain on the electronic VAS without returning to zero during breaks. TSP will be defined as the difference between the mean VAS score from the eight to the tenth stimulus (VAS-II) and the mean VAS value from the first to the fourth stimulus (VAS-I) (e.g., VAS-II minus VAS-I). A higher value indicates enhanced TSP.
Conditioned Pain Modulation | Change from Baseline to after a two-week intervention protocol
  Experimental tonic pain will be evoked on the contralateral leg (at the gastrocnemius muscle) with a continuous cuff-induced painful stimulus, which will be set at 70% of the PTT on that side (conditioning stimulus). Simultaneously, PDT and PTT will be evaluated (test stimulus) on the leg corresponding to the painful/most painful side (NSP group), or the dominant side (control group). The CPM-effect will be defined as the difference between PDT during versus before conditioning. A lower CPM value indicates a less efficient central pain inhibition.
Shoulder Force | Change from Baseline to after a two-week intervention protocol
  The maximal voluntary contraction (MVC) will be measured with a custom built dynamic shoulder dynamometer (Aalborg University, Aalborg, Denmark). Participants will be in a seated upright position with back support and no feet support, and, when required, a corselet will be used to prevent uneven loading of the spine. First, participants will be instructed to raise and lower both shoulders at the same time as much as possible. After that, they will be told to place their shoulders in a relaxed position, and when the pad of the dynamometer is lowered to this level, they will be verbally encouraged to perform a shrug shoulder force in isometric condition for 3 seconds. Recordings will be made twice (2-min break between every test) on the painful shoulder, and the average value will be used for further analysis.
Muscle Stiffness | Change from Baseline to after a two-week intervention protocol
  The biomechanical properties of the upper trapezius will be collected using a handheld myotonometer device, the MyotonPRO, (Myoton AS, Estonia). The MyotonPRO is small, non-invasive, and it has shown good validity and high reliability in larger and smaller body muscles. This device delivers a multi-scan mode of three brief mechanical impulses, each one shortly followed by a quick release, to record the damped natural oscillation of the muscle using an accelerometer.
Muscle Creep | Change from Baseline to after a two-week intervention protocol
  The upper trapezius muscle creep will be collected using a handheld myotonometer device, the MyotonPRO, (Myoton AS, Estonia). The MyotonPRO is small, non-invasive, and it has shown good validity and high reliability in larger and smaller body muscles. This device delivers a multi-scan mode of three brief mechanical impulses, each one shortly followed by a quick release, to record the damped natural oscillation of the muscle using an accelerometer.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Arendt-Nielsen, PhD, Study Director — Aalborg University
Locations (1):
- University of Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided